CLINICAL TRIAL: NCT06067425
Title: A Phase 2, Open-label, Multi-center, 2-stage Sequential Cohort, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Subcutaneous SAR442501 in Pediatric Participants With Achondroplasia
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SAR442501 in Pediatric Participants With Achondroplasia
Acronym: upreACH-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision. Not related to safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DRI16646; U1111-1280-5374 (Registry Identifier: ICTRP); 2023-503677-37 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-09-20; First posted 2023-10-04 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Osteochondrodysplasia
MeSH Terms: conditions — Osteochondrodysplasias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: SAR442501
- Cohort 2 (Experimental)
  Interventions: Drug: SAR442501
- Cohort 3 (Experimental)
  Interventions: Drug: SAR442501

INTERVENTIONS:
Drug: SAR442501 — Solution for injection; Subcutaneous injection

SUMMARY:
This is a Phase 2, open-label, multicenter, study to evaluate safety, tolerability and efficacy of SAR442501 in children from birth up to 12 years of age with Achondroplasia.

DETAILED DESCRIPTION:
Up to approximately 275 weeks: 3 weeks Screening + 52 weeks primary treatment period + up to approximately 216 weeks extended treatment period+ 4 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have ACH with a confirmed mutation in the FGFR3 gene
* Participants and/or parent(s) or legal representative(s) must be willing and able to perform all the study procedures to the best of their physical ability.
* Parent(s) or legal representative(s) capable of giving signed informed consent and participants capable of giving assent when applicable.

Exclusion Criteria:

* Have hypochondroplasia (or the N540K mutation) or short stature condition other than ACH (eg, trisomy 21, pseudochondroplasia)
* Participants have received any dose of medications or investigational product, including human growth hormone, IGF-1, intended to affect participants' stature or body proportions between the completion of OBS16647 and enrollment (Week 0/Day 1/Visit 2).
* Have a history of growth plate closure.
* Long bone fracture within 3 months of enrollment (Week 0/Day 1/Visit 2)
* Current evidence of corneal or retinal disorder/keratopathy.
* Participants have had a previous surgical intervention involving the foramen magnum (Stage 2 only).
* Hyperphosphatemia.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 0 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE), serious adverse events (SAE), and adverse events of special interest (AESI) during the treatment-emergent period | Baseline to Week 52

SECONDARY OUTCOMES:
Change in annualized growth velocity (AGV) Zscore | Baseline to Week 26 and Week 52
Change in AGV (cm/year) | Baseline to Week 26 and Week 52
Change in height Z score | Baseline to Week 26 and Week 52
Change in upper-to-lower body segment ratio | Baseline to Week 26 and Week 52
Change in upper to lower extremity ratio | Baseline to Week 26 and Week 52
Change in sitting to standing height ratio (crown-to-rump length to total length for infants) | Baseline to Week 26 and Week 52
Change in arm span to height ratio | Baseline to Week 26 and Week 52
Change in upper arm to forearm length ratio | Baseline to Week 26 and Week 52
Change in upper leg to lower leg ratio | Baseline to Week 26 and Week 52
Change in head circumference to height ratio | Baseline to Week 26 and Week 52
Change in brainstem parameter | Baseline to Week 52
  Change in surface area of the bony foramen magnum (cm2) as measured by head and neck Magnetic Resonance Imaging (MRI).
Change in skull parameter | Baseline to Week 52
  Change in dimensions of skull base parameters, and degree of synchondroses fusion as measured by head and neck MRI.
Change in spine morphometric parameter | Baseline to Week 52
  Change in grading of cord compression and cord constriction as assessed by head and neck MRI.
Change in volumetric parameter | Baseline to Week 52
  Change in brainstem and spinal cord volume as measured by head and neck MRI.
Change in overall health-related quality of life score in the PedsQL Inventory Generic Core Scale | Baseline to Week 26 and Week 52
  PedsQL Generic Core Scales, global score ranging from 0-100, with higher scores representing better outcomes
Change in fatigue score in the PedsQL Multidimensional Fatigue Scale | Baseline to Week 26 and Week 52
  PedsQL Multidimensional Fatigue Scale, global score ranging from 0-100, with higher scores representing better outcomes
Change in present pain and worst pain rating (PPQ) score | Baseline to Week 26 and Week 52
  Pediatric Pain Questionnaire (PPQ) score value between 0-4. The lower the better.
Change in mobility and symptom rating (STEMS) score | Baseline to Week 26 and Week 52
  Screening Tool for Everyday Mobility and Symptoms (STEMS) score value between 1-5. The lower the better.
Change in developmental score in the Achondroplasia Developmental Recording Form | Baseline to Week 52
  Achondroplasia Developmental Recording Form to record the age at which participants achieve developmental milestones. The earlier the better.
Assessment of pharmacokinetic (PK) parameter: plasma concentration of SAR442501 | Baseline to Week 26 and 52
Assessment of PK parameter: maximum plasma concentration observed (Cmax) | Baseline to Week 26 and 52
Assessment of PK parameter: time to reach Cmax (Tmax) | Baseline to Week 26 and 52
Assessment of PK parameter: Area under the plasma concentration versus time curve calculated using the trapezoidal method during a dose interval (AUC0-t) | Baseline to Week 26 and 52
Assessment of PK parameter: concentration observed before treatment administration during repeated dosing (Ctrough) | Baseline to Week 26 and 52
Assessment of pharmacodynamics (PD) parameter: change in collagen X biomarker (CXM) levels | Baseline to Week 26 and Week 52
Assessment of PD parameter: change in osteocalcin levels | Baseline to Week 26 and Week 52
Assessment of PD parameter: change in bone-specific alkaline phosphatase | Baseline to Week 26 and Week 52
Assessment of PD parameter: change in procollagen type 1 N-terminal propeptide (P1NP) levels | Baseline to Week 26 and Week 52
Assessment of PD parameter: change in collagen-type 1 C-Telopeptide (CTX) levels | Baseline to Week 26 and Week 52
Number of participants with treatment-emergent anti-drug antibodies (ADA) | Baseline to Week 26 and Week 52
Changes in neurological examination | Baseline through Week 26 and Week 52
  Percentage of participants with changes (i.e. abnormal to normal or normal to abnormal) in neurological examination findings

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (9):
- Investigational Site Number : 0360001, Parkville, Victoria, Australia
- China (2):
  - Investigational Site Number : 1560002, Shanghai
  - Investigational Site Number : 1560001, Wuhan
- Italy (2):
  - Investigational Site Number : 3800002, Milan, Lombardy
  - Investigational Site Number : 3800001, Rome, Roma
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (2):
  - Investigational Site Number : 7240002, Vitoria-Gasteiz, Basque Country
  - Investigational Site Number : 7240001, Esplugues de Llobregat, Catalunya [Cataluña]

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org